CLINICAL TRIAL: NCT04271904
Title: Effect of a Sham Anti-inflammatory Diet on Inflammation and Participant Blinding in Spinal Cord Injury: A Pilot Study
Brief Title: Effect of Sham Anti-inflammatory Diet on Inflammation After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AINP001
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injury; Inflammation
MeSH Terms: conditions — Spinal Cord Injuries; Inflammation

STUDY DESIGN:
Intervention Model Description: Eligible participants who consent to study participation will be randomized to one of two groups: placebo diet, or non-dieting control. Those on the placebo diet will be given a meal plan and recipes while the non-dieting control group will be asked to continue eating as usual. The intervention will run for 4-week period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: No other parties will be masked for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Diet (Sham Comparator): Participants on the placebo diet will be given a meal plan and recipes by the study dietitian. The dietitian will assist in developing a diet that is isocaloric to the anti-inflammatory diet and healthy (for the sake of the participants' well-being, and to blind participants), while allowing many foods that are (counterintuitively) pro-inflammatory (e.g. whole wheat bread, white beans, oats, soy, eggplant, raspberries, pumpkin seeds, popcorn, etc). There are many counter-intuitive restrictions in the anti-inflammatory diet that we will be using (banned foods include white beans, soy, eggplant, oats, raspberries, strawberries, prunes, walnuts, cashews, soy milk. Allowed foods include maple syrup, honey, lean beef, lamb, brown rice, feta cheese, butter). Therefore, even fairly astute and educated participants may have trouble discerning which diet they are consuming (anti-inflammatory or placebo).
  Interventions: Other: Placebo Diet
- Non-dieting Control (No Intervention): Those in the non-dieting control condition will not be asked to alter their diet in any way.

INTERVENTIONS:
Other: Placebo Diet — The dietitian will assist in developing a diet that is isocaloric to the anti-inflammatory diet and healthy (for the sake of the participants' well-being, and to blind participants), while allowing many foods that are (counterintuitively) pro-inflammatory (e.g. whole wheat bread, white beans, oats, soy, eggplant, raspberries, pumpkin seeds, popcorn, etc). Occasional "cheat" foods are built into the placebo diet but with more pro-inflammatory options (e.g. two glasses of wine per week).
  Arms: Placebo Diet

SUMMARY:
This pilot study will evaluate the effects of a placebo anti-inflammatory diet in individuals with spinal cord injury. It is being performed to ensure that the placebo diet does not induce reductions in inflammation and also adequately conceals group allocation.

DETAILED DESCRIPTION:
Anti-inflammatory diet is a novel treatment that may be beneficial for managing chronic inflammation and neuropathic pain (NP) after Spinal Cord Injury (SCI). NP is a common complication following SCI that significantly decreases quality of life. Treatment options are limited, and current treatments can have significant side effects. Those with SCI have identified a need for additional treatment options, particularly those that are not medications.

As pain is a subjective outcome, awareness of group allocation could influence treatment expectations and participant rated scores of neuropathic pain. It is therefore important to ensure that an adequate placebo intervention is utilized. This pilot study will assess whether the placebo diet to be used in an upcoming RCT provides sufficient group allocation concealment (i.e. ensure participants are unaware of whether they are on the anti-inflammatory diet or placebo diet). This pilot study will also assess whether the placebo diet is in fact inflammation neutral (ie. induces no reductions in inflammation).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to any study-related activities
2. A spinal cord injury at least 6 months duration, nonprogressive for at least 6 months
3. Dosing of other pain medications (NSAIDs, opioids, non-opioid analgesics, anti-epileptic drugs, antidepressants) should be stable for at least 1 month prior to study entry.

Exclusion Criteria:

1. Current infection of any kind.
2. Presence of other neurologic conditions, medical conditions or pain that could confound the assessment of neuropathic pain after SCI
3. Currently enrolled in another clinical trial
4. Any other significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, may influence the result of the study, or affect the patient's ability to participate in the study
5. Following a physical examination, the patient has any abnormalities that, in the opinion of the investigator would prevent the patient from safe participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein | Baseline and Week-5 (post measures collected following 1-week group allocation period and 4-week intervention)
  Change in plasma C-reactive protein from baseline to post intervention.
Diet Compliance | Week-5 (post measures collected following 1-week group allocation period and 4-week intervention)
  Diet compliance will be assessed following the intervention. Compliance to the specific diet will be assessed by a detailed analysis of all diet records. Each food item will be categorized as either a "food to consume," a "food to avoid," or a "neutral food" based on the parameter of the diet participants who were instructed to follow. Food will also be categorized into servings in accordance with Canada's Food Guide. Therefore, compliance score will be based on standard servings of foods subjects were instructed to eat vs. foods they were instructed to avoid. To account for differences in total energy intake, compliance scores will be expressed as a ratio of the servings of foods to consume over the total servings of food (avoid + consume) multiplied by 100. The percent compliance will then be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Loh, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loh E, Guy SD, Mehta S, Moulin DE, Bryce TN, Middleton JW, Siddall PJ, Hitzig SL, Widerstrom-Noga E, Finnerup NB, Kras-Dupuis A, Casalino A, Craven BC, Lau B, Cote I, Harvey D, O'Connell C, Orenczuk S, Parrent AG, Potter P, Short C, Teasell R, Townson A, Truchon C, Bradbury CL, Wolfe D. The CanPain SCI Clinical Practice Guidelines for Rehabilitation Management of Neuropathic Pain after Spinal Cord: introduction, methodology and recommendation overview. Spinal Cord. 2016 Aug;54 Suppl 1:S1-6. doi: 10.1038/sc.2016.88. PMID 27444714
- [Background] Guy SD, Mehta S, Casalino A, Cote I, Kras-Dupuis A, Moulin DE, Parrent AG, Potter P, Short C, Teasell R, Bradbury CL, Bryce TN, Craven BC, Finnerup NB, Harvey D, Hitzig SL, Lau B, Middleton JW, O'Connell C, Orenczuk S, Siddall PJ, Townson A, Truchon C, Widerstrom-Noga E, Wolfe D, Loh E. The CanPain SCI Clinical Practice Guidelines for Rehabilitation Management of Neuropathic Pain after Spinal Cord: Recommendations for treatment. Spinal Cord. 2016 Aug;54 Suppl 1:S14-23. doi: 10.1038/sc.2016.90. PMID 27444715
- [Background] Allison DJ, Thomas A, Beaudry K, Ditor DS. Targeting inflammation as a treatment modality for neuropathic pain in spinal cord injury: a randomized clinical trial. J Neuroinflammation. 2016 Jun 17;13(1):152. doi: 10.1186/s12974-016-0625-4. PMID 27316678